CLINICAL TRIAL: NCT05293730
Title: Pragmatic Trial of the Impact of the Electronic Frailty Integrated With Social Needs (eFRIEND) on High Cost, High Burden Healthcare Use of Older Adults
Brief Title: Trial of the Impact of the Electronic Frailty Integrated With Social Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00079444
Record Dates: First submitted 2022-03-14; First posted 2022-03-24 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-04

CONDITIONS: Aging
Keywords: Community Health Care Worker; elderly; assistance; at home care
MeSH Terms: conditions — Helping Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Health Worker (CHW)-Led Hybrid In-Person/Telehealth Program Pathway (eFRIEND) (Experimental): Participants in the eFRIEND arm will receive regularly scheduled in-person and telehealth contacts with a CHW.
  Interventions: Behavioral: eFRIEND
- Usual Care (Active Comparator): Usual care group will be monitored passively for outcomes under a waiver of informed consent
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: eFRIEND — eFRIEND is a 6-month CWH-led intervention. All CHW will be part of the research team to ensure successful recruitment and interaction with patients, and all CHW will be certified and have participated in the North Carolina Community Health Worker Standardized Core Competency Training.
  Arms: Community Health Worker (CHW)-Led Hybrid In-Person/Telehealth Program Pathway (eFRIEND)
Other: Usual Care — Routine treatment in primary care
  Arms: Usual Care

SUMMARY:
Participants in Electronic Frailty Integrated with Social Needs (eFRIEND) will randomize to receive regularly scheduled in-person and telehealth contacts with a community health worker (CHW) or continue to receive standard of care. The purpose of this research is to use CHW to help older adults because there may be some resources that could benefit them that they are not aware of or for which they need help applying.

DETAILED DESCRIPTION:
The study team will conduct a pragmatic randomized pilot trial of a CHW-led hybrid in-person/telehealth program pathway (eFRIEND) for frail older adults. Using Zelen's effectiveness design, the study team will identify eligible frail older adults via the Electronic Health Record (EHR). Eligible participants will be randomized to the eFRIEND pathway or usual care. The study team will randomize 2050 older adults (1050 to eFRIEND, 1000 to usual care), with the randomization stratified by primary care clinic. Eligible participants randomized to the eFRIEND pathway will be contacted by phone to discuss study procedures and obtain verbal informed consent. eFRIEND comprises a 6-month intervention. All CHW will be certified and have participated in the North Carolina Community Health Worker Standardized Core Competency Training. CHW are trusted members of the community and are utilized as part of routine care to assist patients. At the first visit, the CHW will assess if the participants have any unmet social and/or functional needs (baseline survey). The frequency and amount of time of each point of contact will be at the discretion of the CHW.

ELIGIBILITY:
Inclusion Criteria:

* Frail based on the electronic Frailty Index (eFI>0.21)
* Live in Forsyth County, NC
* Linked to any Accountable Care Organizations (ACO) registry
* Have a Primary Care Provider (PCP) in Atrium Health Wake Forest Baptist (AHWFB) system, and have seen their PCP or someone else in the clinic of their PCP within the last 12 months

Exclusion Criteria:

* Diagnosis code for dementia in the past 2 years
* Does not speak English

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2050 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2024-05-12 (Actual); Study Completion 2024-05-12 (Actual)

PRIMARY OUTCOMES:
Number of ED Visits or Inpatient Hospitalizations | Month 6
  Healthcare encounters will be tracked using the Electronic Health Record (EHR)
Number of ED Visits or Inpatient Hospitalizations | Month 12
  Healthcare encounters will be tracked using the Electronic Health Record (EHR)

SECONDARY OUTCOMES:
Number of Completed Medicare Annual Wellness Visits (AWVs) | Month 6 and Month 12
  Determined through data extraction from the EHR
Usage of Advance Care Planning (ACP) | Month 6 and Month 12
  Total number of patients who completed ACP based on billing codes (99497 and 99498) from the EHR. The listed billing codes indicate that ACP has been completed at a patient's appointment.
Acceptability of Program | Month 6 and Month 12
  Survey by clinicians at the participating sites. Mean score on the program acceptability survey Acceptability survey is comprised of the Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM). Scores range from 12-60, with higher scores indicating greater acceptability.
Participant Uptake of Home Health Services--Total Number | Month 6 and Month 12
  Care at home survey measuring if patient received home health services with yes or no answer. Total number of participants who say yes.
Participant Uptake of Home Health Services--Proportion | Month 6 and Month 12
  Care at home survey measuring if patient received home health services with yes or no answer. Proportion of participants who say yes.
Proportion of eligible patients who interact with CHW | Month 6 and Month 12
  Shows feasibility of patient recruitment.
Number of Annual Wellness Visits (AWV)s | Month 6 and Month 12
Percentage of Participants who Report Food Insecurity--Total Number | Month 6 and Month 12
  Collected by yes/no response on questionnaire. Subjects who positively report food insecurity are included.
Percentage of Participants who Report Food Insecurity--Proportion | Month 6 and Month 12
  Collected by yes/no response on questionnaire. Subjects who positively report food insecurity are included.
Percentage of Participants who Report Housing Instability--Total Number | Month 6 and Month 12
  Collected by yes/no response on questionnaire. Subjects who positively report housing instability are included.
Percentage of Participants who Report Housing Instability--Proportion | Month 6 and Month 12
  Collected by yes/no response on questionnaire. Subjects who positively report housing instability are included.
Percentage of Participants who Report Lack of Transportation--Total Number | Month 6 and Month 12
  Collected by yes/no response on questionnaire. Subjects who positively report lack of transportation are included.
Percentage of Participants who Report Lack of Transportation--Proportion | Month 6 and Month 12
  Collected by yes/no response on questionnaire. Subjects who positively report lack of transportation are included.
Percentage of Participants who Report Use of Social Services--Total Number | Month 6 and Month 12
  Collected by yes/no response on questionnaire. Subjects who positively report use of social services are included.
Percentage of Participants who Report Use of Social Services--Proportion | Month 6 and Month 12
  Collected by yes/no response on questionnaire. Subjects who positively report use of social services are included.
Percentage of Participants who Report Use of Home Health Services--Total Number | Month 6 and Month 12
  Collected by yes/no response on questionnaire. Subjects who positively report use of home health services are included.
Percentage of Participants who Report Use of Home Health Services--Proportion | Month 6 and Month 12
  Collected by yes/no response on questionnaire. Subjects who positively report use of home health services are included.
Percentage of Participants who Report Social Isolation--Total Number | Month 6 and Month 12
  Collected by yes/no response on questionnaire. Subjects who positively report social isolation are included.
Percentage of Participants who Report Social Isolation--Proportion | Month 6 and Month 12
  Collected by yes/no response on questionnaire. Subjects who positively report social isolation are included.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn E. Callahan, MD, Principal Investigator — Atrium Health Wake Forest Baptist
Locations (1):
- Atrium Health Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Our study, is a Pragmatic Trial of the impact of the Electronic Frailty Integrated with Social Needs (eFRIEND) on high cost, high burden healthcare use of older adults in Atrium Health Wake Forest Baptist, agrees to share study data that fulfill the ICMJE requirements starting after the first 3 months after our study has started and 36 months after our first article publication. We agree to provide data to researchers who can provide our lab with a methodologically sound proposal, and who need our data to help achieve aims outlined in their proposal. The study's data will be comprised of individual participant data that underlie the results reported in our publication. Participant data will be deidentified and can be used in text, tables, figures, and appendices, after approval from the study's primary investigator.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: The requests must include a proposal with clear aims as to why and how the data will be used. If proposal is approved, a data access agreement will need to be signed and will only be accessible for a 36-month period. All requests to gain access to the data will need to be sent to the study's project manager, Renee Woodard, (renee.woodard@wakehealth.edu), with the study's primary investigator copied, Kate Callahan, MD, MS, (kecallah@wakehealth.edu).

DOCUMENTS (1):
  • Informed Consent Form (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT05293730/ICF_000.pdf